CLINICAL TRIAL: NCT02949986
Title: Feasibility of a Tablet-based Fall Prevention Program for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, Courtney D. Hall, Associate Professor, East Tennessee State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETSUIRB0716.5f
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Postural Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tablet-based Fall Prevention (Experimental): The exercise program will be self-administered via a tablet-based version of the fall prevention program and the exercises performed in the home.
  Interventions: Behavioral: Tablet-based Fall Prevention

INTERVENTIONS:
Behavioral: Tablet-based Fall Prevention — The focus of the Otago Exercise Program is on improving strength and balance with a home-based balance exercise program. The program will be self-administered via tablet-based version of the Otago fall prevention program. Participants will complete 2 months of the home-based balance exercise program using the Health in Motion app. Participants will be asked to perform the exercises for 30 minutes 3x/week. Participants will be asked to perform the exercise program for 2 months.

SUMMARY:
There are many exercise approaches that have demonstrated effectiveness in reducing falls and fall risk in community-dwelling older adults. The Otago Exercise Program is one such program. The Otago Exercise Program has been tested in four randomized controlled trials and one controlled multi-center trial and was found to reduce falls in older men and women. The focus of the Otago Exercise Program is on improving strength and balance with a home-based balance exercise program. The goal of the current study is to evaluate whether a self-administered, tablet-based version of the Otago fall prevention program is both feasible and effective for reducing fall risk and improving balance in community-dwelling older adults.

DETAILED DESCRIPTION:
Twenty community-dwelling older adults who satisfy the study criteria will be recruited to participate in this study. This group of participants will be selected to represent the general community-dwelling older adults as much as possible. They will demonstrate a range of ability in terms of their balance and mobility in which some are non-fallers and some fallers. All adults who meet the inclusion/exclusion criteria and have access to the internet via wireless connection will be included.

Participants will be consented for the research study and will be assessed initially, after 1 month of exercise and at the end of 2 months of exercise. Assessment will include questionnaires about health history, including falls, physical activity, balance confidence and system usability. Participants will also complete strength, balance and mobility physical performance tests. Age, sex, presence of comorbidities, medication list, functional abilities, balance confidence, fear of fall behavior and fall history will be assessed by questionnaire. Usability of the tablet-based questionnaire will be assessed by questionnaire. Participants will be tested with standard clinical tests of balance and gait.

Participants will be closely supervised by a Doctor of Physical Therapy (DPT) student during training in how to use the exercise program. Participants will complete a full set of exercises with the tablet in the presence of the DPT student. The DPT student will determine whether participants are safe with the program before allowing them to perform the program on their own at home. If the research team determines that a participant is unable to exercise safely on his/her own he/she will be withdrawn from the study.

The tablet-based, video game exercise program is called Health in Motion and was developed by Blue Marble Game Company. Health in Motion was tested in a pilot study and found to reduce fall risk in 8 of 15 older participants without any adverse events. Participants will complete 2 months of the home-based balance exercise program using the Health in Motion app. Participants will be asked to perform the exercises for 30 minutes 3x/week. Participants will be asked to perform the exercise program for 2 months.

Performance scores from the clinical gait and balance measures obtained during the initial visit will be compared to the performance scores obtained after 1 month and 2 months of performing the exercise program. We hypothesize that balance and gait will improve following 2 months of performing the tablet-based fall prevention exercise program at home. The assessments performed by the DPT students and by the participant using the app will be compared. We hypothesize that the scores from self-assessment will closely correlate to the students' assessment. The system usability score will be examined to understand issues associated with using technology. We hypothesize that older adults will enjoy performing the exercises using the tablet format.

ELIGIBILITY:
Inclusion Criteria:

* age at least 60 years, ability to ambulate household distance without an assistive device; and ability to stand independently for twenty minutes

Exclusion Criteria:

* cognitive impairment (based on Mini Mental Status Exam), unstable medical condition, progressive neurological condition, severe pain with weight bearing, and severe vision impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Activity-specific balance confidence (ABC) | 2 months
  ABC is a 16-item questionnaire regarding confidence to perform different activities (e.g., walking around the house, up and down stairs, and on icy surfaces) without losing balance. The scale ranges from 0% (no confidence at all) to 100% (completely confident). An overall average balance confidence score will be calculated for each subject.

SECONDARY OUTCOMES:
Timed up and go test (TUG) | 2 months
  The timed up and go test (TUG) is commonly used to assess functional mobility in older adults and is sensitive to fall risk (Shumway-Cook et al., 2000). The test involves standing up, walking as quickly and safely as possible for 3 m, turning around, walking back and then sitting down. Time to complete the TUG will be recorded.
Functional Gait Assessment (FGA) | 2 months
  The 10 items of the FGA include walking while changing speed and turning the head, walking over obstacles, walking tandem, backward and with eyes closed and stair climbing. A maximum total score of 30 is possible with scores < 22 indicating high risk for falling (Wrisley et al., 2010).
Preferred gait speed | 2 months
  Gait speed will be determined by instructing participants to walk at their normal pace over a 9-m pathway. The time to walk the middle 6 m will be measured using a stopwatch and gait speed calculated. Gait speed has excellent test-retest reliability (r = 0.90; Bohannon, 1997) and slower gait speed is associated with fall risk (Montero-Odasso et al., 2005).
Single Leg Stance Test | 2 months
  The Single Leg Stance Test is a test of balance and requires participants to stand on one leg for up to 30 seconds. Up to three trials, using each leg will be performed. SLS is correlated with injurious falls (Vellas et al., 1997).
Modified clinical test of sensory interaction on balance (mCTSIB) | 2 months
  The mCTSIB is organized into a series of 4 conditions of increasing difficulty and timed for a maximum of 30 seconds for each condition. The first two conditions involve a stable support surface with eyes open and eyes closed. The last two conditions involve a foam surface with eyes open and eyes closed. The mCTSIB score is the sum of the average time for each condition.
Physical Activity Scale for the Elderly (PASE) | 2 months
  The PASE is comprised of self-reported occupational, household and leisure items over a one-week period and can be administered by telephone, mail or in-person.
Fear of Falling Avoidance Behavior Questionnaire | 2 months
  The Fear of Falling Avoidance Behavior Questionnaire is a 14 item questionnaire that measures avoidance of behaviors due to fear of falling (Landers, Durand, Powell, Dibble, Young, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Hall, PhD, Principal Investigator — East Tennessee State University
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No